CLINICAL TRIAL: NCT01834612
Title: Clinical Evaluation of the Zynex Blood Volume Monitor (CM1500) in Healthy Adult Volunteers During a Blood Draw
Brief Title: Evaluation of the Zynex Blood Volume Monitor in Healthy Adult Volunteers During a Blood Draw
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zynex Monitoring Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Zynex 750
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Blood Loss
Keywords: blood loss, hemorrhage, hemorrhagic shcok
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blood draw (Active Comparator): CM1500 with blood draw
  Interventions: Device: CM1500
- No blood draw (Sham Comparator): CM 1500 with no blood draw
  Interventions: Device: CM1500

INTERVENTIONS:
Device: CM1500 — blood volume monitor

SUMMARY:
To determine if a manual blood loss can be detected using the non-invasive blood monitor.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer
* between 18 to 50 years of age
* weight between 157 to 220 lbs

Exclusion Criteria:

* unstable or untreated cardia disease
* alcohol consumption in 24 hours prior to screening
* tobacco use in 4 hours prior to screening
* pregnancy
* infection
* Hemoglobin < 12.5 g/dL at time of procedure

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2013-03-11 (Actual); Study Completion 2013-03-11 (Actual)

PRIMARY OUTCOMES:
Detect change in blood volume by non-invasive monitoring during whole blood draw | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Chris Galloway, MD, Principal Investigator — Davita Clinical Research
Locations (1):
- DaVita Clinical Research, Lakewood, Colorado, United States